CLINICAL TRIAL: NCT00770341
Title: A Phase III Randomized, Open-labeled Clinical Trial of MK-3009 (Daptomycin) in Patients With Skin and Soft Tissue Infections, Septicemia and Right-sided Infective Endocarditis Caused by MRSA
Brief Title: A Study of MK-3009 in Japanese Patients With Skin or Blood Stream Infections Caused by Methicillin-resistant Staphylococcus Aureus (MK-3009-002)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3009-002; 2008_564
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Staphylococcal Infection
MeSH Terms: conditions — Staphylococcal Infections | interventions — Daptomycin

ARMS (3):
- MK-3009 (daptomycin) 4 mg/kg (Experimental)
  Interventions: Drug: Daptomycin 4 mg/kg
- Vancomycin (Active Comparator)
  Interventions: Drug: Comparator: vancomycin
- MK-3009 (daptomycin) 6 mg/kg (Experimental)
  Interventions: Drug: Daptomycin 6 mg/kg

INTERVENTIONS:
Drug: Daptomycin 4 mg/kg — MK3009 (daptomycin) once daily by intravenous (IV) drip, 4 mg/kg for 7-14 days for skin and soft tissue infections (SSTI)
  Other Names: MK3009
  Arms: MK-3009 (daptomycin) 4 mg/kg
Drug: Comparator: vancomycin — vancomycin 1g, twice daily (b.i.d.) by IV drip, for 7-14 days
  Arms: Vancomycin
Drug: Daptomycin 6 mg/kg — MK-3009 (daptomycin) once daily by intravenous drip, 6 mg/kg for 14-42 days for septicemia or right-sided infective endocarditis
  Arms: MK-3009 (daptomycin) 6 mg/kg

SUMMARY:
The study investigates the efficacy and safety of MK-3009 in participants with skin infections, septicemia and right-sided infective endocarditis (RIE) caused by methicillin-resistant Staphylococcus aureus (MRSA).

ELIGIBILITY:
Inclusion Criteria:

* Both Sexes, Aged 20 Years Or Older
* Japanese Participants With Skin And Soft Tissue Infections, Septicemia, or RIE Known Or Suspected To Be Caused By MRSA
* Written Informed Consent

Exclusion Criteria:

* Participants With Skin and Soft Tissue infections That Can Be Treated By Surgery Alone
* Participants With Pneumonia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2008-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Aikawa N, Kusachi S, Mikamo H, Takesue Y, Watanabe S, Tanaka Y, Morita A, Tsumori K, Kato Y, Yoshinari T. Efficacy and safety of intravenous daptomycin in Japanese patients with skin and soft tissue infections. J Infect Chemother. 2013 Jun;19(3):447-55. doi: 10.1007/s10156-012-0501-9. Epub 2012 Oct 20. PMID 23085743
- [Derived] Takesue Y, Mikamo H, Kusachi S, Watanabe S, Takahashi K, Yoshinari T, Ishii M, Aikawa N. Correlation between pharmacokinetic/pharmacodynamic indices and clinical outcomes in Japanese patients with skin and soft tissue infections treated with daptomycin: analysis of a phase III study. Diagn Microbiol Infect Dis. 2015 Sep;83(1):77-81. doi: 10.1016/j.diagmicrobio.2015.05.013. Epub 2015 May 28. PMID 26072149

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-3009 (Daptomycin) 4 mg/kg: Intravenous (IV) Daptomycin 4 mg/kg once daily for skin & soft tissue infections (SSTI)
- Vancomycin: IV Vancomycin 1 g twice daily for SSTI
- MK-3009 (Daptomycin) 6 mg/kg: IV Daptomycin 6 mg/kg once daily for Septicemia and right-sided infective endocarditis (RIE)
Period: Overall Study
Arm/Group | MK-3009 (Daptomycin) 4 mg/kg | Vancomycin | MK-3009 (Daptomycin) 6 mg/kg
Started | 89 (Number randomized) | 22 (Number randomized) | 11 (Number randomized)
Completed | 77 | 17 | 8
Not Completed | 12 | 5 | 3
Not completed — Did not meet eligibility criteria | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Clinical Adverse Event | 3 | 1 | 2
Not completed — Laboratory adverse event | 3 | 3 | 0
Not completed — Lack of Efficacy | 3 | 0 | 1
Not completed — Other | 1 | 0 | 0
Not completed — Not treated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-3009 (Daptomycin) 4 mg/kg | Vancomycin | MK-3009 (Daptomycin) 6 mg/kg | Total
Number analyzed (Participants) | 88 | 22 | 11 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] — Age information was for all treated participants (N=121)
  years | 65.6 (16.0) | 61.7 (17.1) | 77.7 (10.9) | 66.0 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 7 | 9 | 57
  Male | 47 | 15 | 2 | 64
Region of Enrollment [Number; unit: participants]
  Japan | 88 | 22 | 11 | 121

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Adjudication Committee (EAC) Assessment of Number of Participants With Clinical Success at Test of Cure (TOC)
Description: Clinical Success = Study investigator's Clinical Response confirmed by the EAC as either cured or improved at end of treatment (EOT).
  MITT-MRSA (modified intent-to-treat - methicillin-resistant Staphylococcus aureus) was a subset of allocated participants with participants who were excluded for any of the following reasons: no MRSA isolated + any 1 of the following: failure to receive ≥1 dose of study drug, lack of all post-allocation primary and secondary endpoint data after ≥1 dose of study drug, no gram (+) coccus isolated at baseline.
Time Frame: 7-14 days for SSTI, 14-42 days for septicemia and right-sided infective endocarditis (RIE)
Population: MITT-MRSA; One participant with possible MRSA RIE was enrolled. This participant was excluded from the efficacy population.
Measure: Number; unit: Participants
Arm/Group | MK-3009 (Daptomycin) 4 mg/kg | Vancomycin | MK-3009 (Daptomycin) 6 mg/kg
Number analyzed (Participants) | 55 | 19 | 4
Participants | 45 | 16 | 2

2. Secondary Outcome: EAC Assessment of Number of Participants With Clinical Success at End of Treatment (EOT).
Description: Clinical Success = Study investigator's Clinical Response confirmed by the EAC as either cured or improved at EOT.
Time Frame: 7-14 days for SSTI, 14-42 days for septicemia and RIE
Population: MITT-MRSA; one participant with possible MRSA RIE was enrolled into this study. This participant was excluded from the efficacy population.
Measure: Number; unit: Participants
Arm/Group | MK-3009 (Daptomycin) 4 mg/kg | Vancomycin | MK-3009 (Daptomycin) 6 mg/kg
Number analyzed (Participants) | 54 | 19 | 4
Participants | 46 | 16 | 2

3. Primary Outcome: Efficacy Adjudication Committee (EAC) Assessment of Number of Participants With Microbiological Response at TOC
Description: Response = eradicated or presumed eradicated.
  Eradicated was defined as absence of the admission pathogen in a culture obtained in the absence of potentially effective antibiotics for the pathogen.
  Presumed eradicated was defined as no material for culture was available due to improvement of infection, but the admission pathogen was presumed to be eradicated because the participant was deemed "Cured" or "Improved" by the investigator and the participant did not receive potentially effective antibiotics for the pathogen.
Time Frame: 7-14 days for SSTI, 14-42 days for septicemia and RIE
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | MK-3009 (Daptomycin) 4 mg/kg | Vancomycin | MK-3009 (Daptomycin) 6 mg/kg
Number analyzed (Participants) | 55 | 19 | 4
Participants | 31 | 9 | 2

4. Secondary Outcome: EAC Assessment of Number of Participants With Microbiological Response at End of Treatment (EOT).
Description: as for outcome 3
Time Frame: 7-14 days for SSTI, 14-42 days for septicemia and RIE
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | MK-3009 (Daptomycin) 4 mg/kg | Vancomycin | MK-3009 (Daptomycin) 6 mg/kg
Number analyzed (Participants) | 55 | 19 | 4
Participants | 24 | 9 | 4

5. Secondary Outcome: Study Investigators' Assessment of Clinical Response at EOT
Description: Clinical Success = Study investigator's Clinical Response confirmed by the EAC as either cured or improved at EOT.
Time Frame: 7-14 days for SSTI, 14-42 days for septicemia and RIE
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | MK-3009 (Daptomycin) 4 mg/kg | Vancomycin | MK-3009 (Daptomycin) 6 mg/kg
Number analyzed (Participants) | 54 | 19 | 4
Participants | 47 | 18 | 3

6. Secondary Outcome: Study Investigators' Assessment of Clinical Response at TOC
Description: Clinical Success = Study investigator's Clinical Response confirmed by the EAC as either cured or improved at EOT.
Time Frame: 7-14 days for SSTI, 14-42 days for septicemia and RIE
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | MK-3009 (Daptomycin) 4 mg/kg | Vancomycin | MK-3009 (Daptomycin) 6 mg/kg
Number analyzed (Participants) | 55 | 19 | 4
Participants | 48 | 17 | 2

ADVERSE EVENTS:
Arm/Group | NOT TREATED | DAPTOMYCIN (4 MG/KG) | VANCOMYCIN | DAPTOMYCIN (6 MG/KG)
Serious Adverse Events (participants affected / at risk) | 0/1 | 6/88 | 4/22 | 4/11
Other Adverse Events (participants affected / at risk) | 0/1 | 34/88 | 11/22 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOT TREATED (N=1) | DAPTOMYCIN (4 MG/KG) (N=88) | VANCOMYCIN (N=22) | DAPTOMYCIN (6 MG/KG) (N=11)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTRA-ABDOMINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANAPHYLACTIC SHOCK (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SKELETAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM ST SEGMENT DEPRESSION (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOPHARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOT TREATED (N=1) | DAPTOMYCIN (4 MG/KG) (N=88) | VANCOMYCIN (N=22) | DAPTOMYCIN (6 MG/KG) (N=11)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (3) | 1 (1)
GASTRIC VOLVULUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERITONITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PAIN (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 6 (6) | 2 (2) | 0 (0)
ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARTHRITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CATHETER RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
JOINT ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCLE ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 9 (9) | 3 (3) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 9 (9) | 3 (3) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BLOOD POTASSIUM INCREASED (Investigations) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
BLOOD URINE PRESENT (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
EOSINOPHIL COUNT INCREASED (Investigations) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
GLUCOSE URINE PRESENT (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
ANGIOPATHY (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.